CLINICAL TRIAL: NCT02919709
Title: Follow up of Patients With Aortic Aneurysm by Dosage of Circulant Endothelial Progenitor Cells
Acronym: ANOPEC 3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P/2013/186
Record Dates: First submitted 2016-09-27; First posted 2016-09-29 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Thoracic or Abdominal Aortic Aneurysm With no Indication for Surgical Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- thoracic or abdominal aortic aneurysm (Experimental)
  Interventions: Biological: blood taking

INTERVENTIONS:
Biological: blood taking

SUMMARY:
The study aims to investigate the existence of a reliable correlation between the progression of aortic diameters and blood levels of circulant endothelial progenitor cells CD34+ in patients with not surgical aortic aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 or more.
2. Patients diagnosed with a thoracic or abdominal aortic aneurysm with no indication for surgical treatment (diameters > 30 mm but < 50 mm).
3. Patients accepting to sign a specific informed consent.

Exclusion Criteria:

1. Unstable coronary artery disease.
2. Congenital heart disease.
3. Any evolving infectious syndrome or viral infection (HIV, HBV or HCV).
4. Any chronic inflammatory or autoimmune disease.
5. Prior administration of G-CSF; EPO; GM-CSF.
6. Liver failure.
7. Prior oncologic disease or ongoing cancer with a life expectancy < 1 year.
8. Dementia.
9. Pregnancy.
10. Patients aged < 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
progenitor cells CD34+ blood levels | At diagnosis of aneurysm
progenitor cells CD34+ blood levels | 6 month after disgnosis
progenitor cells CD34+ blood levels | 12 month after diagnosis
progenitor cells CD34+ blood levels | 18 month after diagnosis
progenitor cells CD34+ blood levels | 24 month after diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No